CLINICAL TRIAL: NCT02146287
Title: Preterm Infants: Light Effects on Health and Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00011520; R01NR008044 (NIH)
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Preterm Infant Health; Preterm Infant Development
Keywords: cycled light; preterm infants; infant neurodevelopment; infant sleep

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Cycled Light (Active Comparator): Infants received day night cycling of light on a 12-hour on and 12-hour off basis beginning at 28 weeks PMA
  Interventions: Other: Cycled Light
- Late Cycled Light (Active Comparator): Infants received day night cycling of light on a 12-hour on and 12-hour off basis beginning at 36 weeks PMA
  Interventions: Other: Cycled Light

INTERVENTIONS:
Other: Cycled Light — Cycled light was provided in an 11-hour-on, 11-hour-off pattern. Daylight (240-700 lux) was provided with the incubator cover folded on top of the incubator allowing light in from four sides, or with the bassinet cover off during day hours (0730-1830). With the daylight range of 240-700 lux and limited access to natural light, excessive daylight was prevented.
  Continuous near darkness was provided as (5-30 lux) throughout the day except from 0630-0730 and 1830-1930, when lighting levels varied based on nursing care needs at the change of shift. Near-darkness (5-30 lux) was provided by using incubator (totally covered or with the front flap back) and bassinet covers, and dimming individual bedside light during the day (0730-1830) and night hours (1930-0630).

SUMMARY:
Preterm babies cared for in the intensive care nursery are exposed to amounts of light that are very different from the exposures to an unborn baby or the newborn term baby. Currently many nurseries try to protect premature babies from too much light. They may also try to create light conditions of day and night like many parent homes. Some studies have shown improvements in health and development of babies cared for in nurseries that try to change light for premature babies.

ELIGIBILITY:
Inclusion Criteria:

* Infants were < 7 days of age and were born at 28 weeks or < 28 weeks

Exclusion Criteria:

* known anomalies associated with neurological or visual problems (e.g., congenital glaucoma, Down Syndrome)

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2003-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Infant weight gain trajectory | weekly inpatient up to 52 weeks post menstral age (PMA) and at outpatient visits to 18 months
  This measure was single blinded.
Change in sleep development during hospitalization | Every three weeks up to 52 weeks PMA
  Change in the developmental pattern of four sleep wake states (active, quiet, transition, awake) were evaluated during hospitalization.
Change in sleep development after discharge home | Every 5 months following hospital discharge up to 24 months PMA
  Change in the development of sleep and wake bouts were evaluated following hospital discharge until the infant reached 24 months PMA
Mental Development | 9 months PMA
  Mental development was measured using the Bayley Scales of Infant Development.
Psychomotor Development | 9 months PMA
  Psychomotor Development was measured using the Bayley Scales of Infant Development
Mental Development | 18 months PMA
  Mental development was measured using the Bayley Scales of Infant Development.
Psychomotor Development | 18 months PMA
  Psychomotor Development was measured using the Bayley Scales of Infant Development

SECONDARY OUTCOMES:
Length of Hospitalization in Days | At hospital discharge from 0 to 222 days
  Length of hospitalization from birth until discharge home.
Severity of Retinopathy of Prematurity (ROP) | Up to 52 weeks
  ROP change over time and degree of severity was assessed until 24 months PMA
visual acuity | Measures at 12 months PMA
Neurological development | 9 months PMA
  Neurological development was assessed by a neurological exam as either normal, suspect or abnormal and the presence of absence of Cerebral Palsy
Brainstorm Auditory Evoked Potentials | 6 months
Neurological development | 18 months PMA
  Neurological development was assessed by a neurological exam as either normal, suspect or abnormal and the presence of absence of Cerebral Palsy
Change in Retinopathy of Prematurity (ROP) | Every two weeks during hospitalization after 30 weeks PMA up to 52 weeks PMA and during outpatient visits up to 24 months PMA
  ROP change over time and degree of severity was assessed until 24 months PMA

CONTACTS AND LOCATIONS:
Overall Officials: Debra H Brandon, PhD, Principal Investigator — Duke University School of Nursing

REFERENCES:
- [Derived] Morag I, Xiao YT, Bruschettini M. Cycled light in the intensive care unit for preterm and low birth weight infants. Cochrane Database Syst Rev. 2024 Dec 19;12(12):CD006982. doi: 10.1002/14651858.CD006982.pub5. PMID 39699174
- [Derived] Park J, Knafl G, Thoyre S, Brandon D. Factors associated with feeding progression in extremely preterm infants. Nurs Res. 2015 May-Jun;64(3):159-67. doi: 10.1097/NNR.0000000000000093. PMID 25932696